CLINICAL TRIAL: NCT04011566
Title: Assessment of ShuntCheck Performance Characteristics in Asymptomatic Patients With Normal Pressure Hydrocephalus
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University of South Florida (Other)
Collaborators: NeuroDx Development (Industry)
Responsible Party: Principal Investigator, Naomi Abel, Assistant Professor, College of Medicine Neurosurgery, University of South Florida
Other Study IDs: Pro00040697
Record Dates: First submitted 2019-06-18; First posted 2019-07-08 (Actual); Last update posted 2022-09-30 (Actual); Status verified 2022-09

CONDITIONS: Hydrocephalus, Normal Pressure
Keywords: Asymptomatic Normal Pressure Hydrocephalus; Ventriculoperitoneal Shunt
MeSH Terms: conditions — Hydrocephalus, Normal Pressure

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- ShuntCheck: Participants will be administered the ShuntCheck diagnostic test.
  Interventions: Diagnostic Test: ShuntCheck

INTERVENTIONS:
Diagnostic Test: ShuntCheck — The intervention is an FDA-cleared device utilizing a transcutaneous thermal convection to analyze shunt flow.

SUMMARY:
The purpose of the study is to determine if the ShuntCheck test can correctly identify flow or no flow in a ventriculoperitoneal shunt in patients with asymptomatic normal pressure hydrocephalus.

ELIGIBILITY:
Inclusion Criteria:

* Asymptomatic men or women 40 years old or older and have a ventriculoperitoneal shunt placed for normal pressure hydrocephalus and are visiting for routine care.
* Capable of providing valid signed informed consent, or has a legal guardian, health care agent, or surrogate decision maker capable of providing valid, signed informed consent.

Exclusion Criteria:

* Presence of multiple shunts, or presence of more than one distal shunt catheter (regardless of function) crossing the clavicle ipsilateral to the shunt with suspected obstruction;
* ShuntCheck test would interfere with standard patient care, or emergency shunt surgery that cannot be delayed is indicated;
* Presence of an interfering open wound or edema over any portion of the ventriculoperitoneal shunt.

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population will consist of asymptomatic normal pressure hydrocephalus research subjects who have a ventriculoperitoneal shunt with a single ventricular catheter implanted for adult hydrocephalus and are visiting for routine care. Evaluation will be within 2 weeks of shunt placement.
Sampling Method: Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2019-06-11 (Actual); Primary Completion 2024-06 (Estimated); Study Completion 2025-01 (Estimated)

PRIMARY OUTCOMES:
Specificity of ShuntCheck test | 15 minutes
Negative Predictive Value of ShuntCheck test | 15 minutes

SECONDARY OUTCOMES:
Specificity of performing ShuntCheck test twice | 60 minutes
Negative Predictive Value of performing ShuntCheck test twice | 60 minutes

CONTACTS AND LOCATIONS:
Overall Officials: Naomi Abel, MD, Principal Investigator — University of South Florida
Locations (1):
- University of South Florida Department of Neurological Surgery and Brain Repair, Tampa, Florida, United States

IPD SHARING:
Plan to Share IPD: Yes
individual participant data that underlies the results reported after deidentification and statistical analysis will be shared following publication for 5 years with researchers who provide a methodologically sound proposal
Supporting Information: CSR
Time Frame: individual participant data that underlies the results reported after deidentification and statistical analysis will be shared following publication for 5 years with researchers who provide a methodologically sound proposal
Access Criteria: data use agreement required and methodologically sound proposal